CLINICAL TRIAL: NCT06887478
Title: Examination of Balance-Gait Parameters and Fall Effect of Flexor Hallucis Longus Muscle Strengthening Training in Geriatric Group
Brief Title: Flexor Hallucis Longus Training and Balance-Gait in Geriatrics
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lokman Hekim University (Other Government)
Responsible Party: Principal Investigator, Hüseyin Gerdan, PhD thesis student, Lokman Hekim University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024049
Record Dates: First submitted 2025-03-08; First posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Flexor Hallucis Longus Muscle Strength in Elderly Individuals
Keywords: elderly; flexor hallucis longus; balance; gait; falls
MeSH Terms: interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Physiotherapist-Assisted Isolated FHL Strengthening Exercise Group (Experimental): The intervention for the "Physiotherapist-Assisted Isolated FHL Strengthening Exercise Group (FHL-SET)" will consist of physiotherapist-guided, isolated strengthening exercises specifically targeting the Flexor Hallucis Longus (FHL) muscle. Participants will engage in exercises designed to isolate and strengthen the FHL muscle through controlled and progressive resistance. Sessions will occur three times a week for 8 weeks, with the physiotherapist providing individualized adjustments and ensuring proper technique and progression.
  Interventions: Other: Exercise
- Home-Based Foot and Ankle Strengthening Exercise Training Group (Experimental): After the initial assessments, the participants in this group will receive home-based foot and ankle strengthening exercises three times a week for 8 weeks. They will be monitored weekly using an exercise log. The Home-Based Exercise Group (EvT-KE) will be taught general foot exercises without progression in resistance. These exercises include ankle rotations, toe raises, toe lifts, rolling a ball under the foot for 2 minutes, picking up marbles with toes, towel collection exercises, and foot shortening exercises.
  Interventions: Other: Exercise
- Control Group (No Intervention): For the Control Group, initial and final assessments will be conducted at the beginning of the study and at the end of 8 weeks. No exercise program will be provided during this period. After the study, necessary exercises and recommendations will be given.

INTERVENTIONS:
Other: Exercise — A progressive resistance exercise program focusing on strengthening the flexor hallucis longus (FHL) muscle in elderly participants.
  Arms: Home-Based Foot and Ankle Strengthening Exercise Training Group; Physiotherapist-Assisted Isolated FHL Strengthening Exercise Group

SUMMARY:
Examination of Balance-Gait Parameters and Fall Effect of Flexor Hallucis Longus Muscle Strengthening Training in Geriatric Group It has been demonstrated that the reduction in the strength of the toe flexor muscles is an independent indicator of falls in geriatric individuals. However, the extent of this strength loss and the effects of strengthening training programs on balance, gait parameters, and falls are not well understood.

Objective: The aim is to investigate whether a progressive resistance exercise program, focusing specifically on the flexor hallucis longus (FHL) muscle, can improve toe flexor strength and influence gait, balance, and falls in geriatric individuals.

Materials and Methods: Individuals over the age of 65 who are willing to participate in the study will be included. The participants will be divided into three groups: individual exercise group, home exercise group, and control group. Individuals who are unable to walk independently, have severe musculoskeletal disorders, have hallux rigidus deformity, suffer from orthostatic hypotension, have difficulty understanding instructions, or have diabetic neuropathy will be excluded from the study. After obtaining socio-demographic information from the participants, anthropometric measurements will be taken. Toe grip strength will be assessed using a digital dynamometer, and the strength of the intrinsic foot muscles and lower extremity antigravity muscles will also be measured using a digital dynamometer. Balance parameters will be evaluated using the Berg Balance Scale, Functional Reach Test, Timed Up and Go Test, while gait parameters will be assessed using the 10-meter walk test and Tinetti Gait Scale. Fall parameters will be assessed by the Falls Efficacy Scale and fall frequency.

The collected data will be analyzed using SPSS (Statistical Package for Social Sciences) software.

ELIGIBILITY:
Inclusion Criteria:

* Individuals over the age of 65,
* Individuals who do not have hearing or speech problems,
* Individuals who do not have any neurological, orthopedic or visual problems that would prevent walking (can walk 10 meters independently)
* Individuals who score 24 points and above in the Mini Mental Test evaluation.

Exclusion Criteria:

* Those who cannot walk independently,
* Those with serious musculoskeletal system disorders,
* Those with hallux rigidus deformity,
* Those with orthostatic hypotension,
* Those who have difficulty understanding instructions and those with diabetic neuropathy.

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Gender Based: Yes — over 65 years old
Enrollment: 66 (Estimated)
Dates: Start 2025-01-10 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-04-01 (Estimated)

PRIMARY OUTCOMES:
Muscle Strength Measurement | pre-intervention, immediately after the intervention
  Flexor hallucis longus strength and toe grip strength will be assessed using Dynamo by Vald branded dynamometer. The results will be reported in Newtons.
balance assessment | pre-intervention, immediately after the intervention
  berg balance scale
gait | pre-intervention, immediately after the intervention
  gait speed, cadence

CONTACTS AND LOCATIONS:
Locations (1):
- Atakum Nursing Home, Elderly Care and Rehabilitation Center, Samsun, Samsun, Turkey (Türkiye)